CLINICAL TRIAL: NCT02020408
Title: Monoamine Contributions to Neurocircuitry in Eating Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Walter Kaye, MD, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 090661; R01MH092793 (NIH)
Record Dates: First submitted 2013-12-11; First posted 2013-12-24 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2019-12

CONDITIONS: Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Raclopride; 3-amino-4-(2-dimethylaminomethylphenylsulfanyl)benzonitrile; Amphetamine; Dextroamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [11C]raclopride, [11C]DASB, amphetamine (Experimental): One time administration of oral amphetamine based on subject's weight (0.5 mg/kg). One PET scan using [11C]DASB. Two PET scans using [11C]raclopride.
  Interventions: Drug: [11C]raclopride; Drug: [11C]DASB; Drug: amphetamine

INTERVENTIONS:
Drug: [11C]raclopride — 1.[11C]raclopride -The change (Δ) in BPND (the difference between the [11C]raclopride BPND at baseline and post-AMPH treatment normalized to the baseline BPND
  Other Names: Raclopride, serial number 009
Drug: [11C]DASB — BPND of [11C]DASB.
  Other Names: DASB, serial number 0011
Drug: amphetamine — The change (Δ) in BPND (the difference between the [11C]raclopride BPND at baseline and post-AMPH treatment normalized to the baseline BPND.
  Other Names: dextroamphetamine

SUMMARY:
This study will use brain imaging technologies to measure several neurotransmitters (serotonin and dopamine) that contribute to our abilities to respond to reward or inhibit our impulses, and which are known to be altered in the brain of people with anorexia nervosa (AN) and bulimia nervosa (BN). Because palatable food stimulates dopamine secretion, we propose to use a challenge with brain imaging that will stimulate dopamine release which we hypothesize will generate anxiety rather than pleasure in AN, and will help explain why AN restrict eating in order to reduce anxiety. This study will help to understand the unique puzzling symptoms in eating disorders and contribute to finding better methods for identifying effective treatments for these often relapsing and sometimes chronic disorders.

DETAILED DESCRIPTION:
Alterations of serotonin (5-HT) and dopamine (DA) activity may contribute to extremes of appetitive behaviours in anorexia nervosa (AN) and bulimia nervosa (BN), through effects on inhibitory and reward neural pathways. To avoid the confounding effects of malnutrition, and because they have behaviours and neural circuit alterations relevant for this study, we will study 25 recovered (REC) restricting-type AN, 25 REC bulimic-type AN (AN-BN), 25 REC BN, and 25 control women (CW). This 5 year study, of women 18 to 45 years old, will employ positron emission tomography (PET) imaging with radioligands for the 5-HT transporter ([11C]DASB) and DA D2/D3 receptors ([11C]raclopride).

ELIGIBILITY:
Inclusion

* history of Diagnostic and Statistical Manual (DSM-IV) diagnosis of anorexia or bulimia.
* AN women have history of average body weight (ABW) below 85% for height.
* AN-BN subjects have history of ABW below 85% ABW.
* AN-BN subjects have history of binging/purging behaviors during a period of low weight.
* Subjects must be right-handed.
* Subjects have been recovered for 12 months or more.

Exclusion

* Diagnosis of alcohol or drug abuse or dependence in the 3 months.
* Alcohol or substance use within 30 days.
* Current diagnosis of an Axis I disorder.
* Organic brain syndromes, dementia, psychotic disorders, or mental retardation.
* Neurological or medical disorders such as seizure disorder, renal disease, diabetes, thyroid disease, EKG indicative of electrolyte imbalance
* BN subjects whose purging methods were the use of laxatives, diuretics
* Use of psychoactive medication in the 3 months.
* Pregnancy or lactation.
* Tobacco use in the 3 months.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-05; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kaye, MD, Principal Investigator — UCSD; Ursula Bailer, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- [11C]Raclopride, [11C]DASB, Amphetamine: 1. healthy control women (CW);
  2. women recovered from restricting type anorexia nervosa (REC AN);
  3. women recovered from bulimic type anorexia nervosa (REC AN-BN)
  4. women recovered from from bulimia nervosa (REC BN)
Period: Overall Study
Arm/Group | [11C]Raclopride, [11C]DASB, Amphetamine
Started | 88
Completed | 85
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: According to the study protocol and inclusion criteria all participants needed to be female, between age 18 and 65 and were enrolled in the US.
Arm/Group | [11C]Raclopride, [11C]DASB, Amphetamine
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 72
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: 5-HT Transporter Binding as Measured During the PET Scan
Description: Use PET and [11C]DASB to explore 5-HTT receptor binding potential midbrain and striatal regions of interest in eating disorder subtypes.
  The Binding Potential (BP) was calculated as BP Non Displaceable (ND) = (VT/VND) -1. [VT = distribution volume in tissue; VND = non-displaceable distribution volume]. The binding of the 5-HTT on PET presumably reflects 5-HTT density and/or affinity.
Time Frame: 90 minute PET scan
Measure: Mean (Standard Deviation); unit: binding potential (BPND)
Groups:
- [11C]DASB Binding Potential Control Women: [11C] DASB Binding potential (BPND) in control women (healthy controls)
- [11C]DASB Binding Potential in REC AN: [11C]DASB binding potential in women recovered from restricting type anorexia nervosa (REC AN)
- [11C]DASB Binding Potential in REC ANBN: [11C]DASB binding potential in women recovered from bulimic type anorexia nervosa (REC AN-BN)
- [11C]DASB Binding Potential in REC BN: [11C]DASB binding potential in women recovered from bulimia nervosa (REC BN)
Arm/Group | [11C]DASB Binding Potential Control Women | [11C]DASB Binding Potential in REC AN | [11C]DASB Binding Potential in REC ANBN | [11C]DASB Binding Potential in REC BN
Number analyzed (Participants) | 24 | 18 | 16 | 8
binding potential (BPND)
  [11C]DASB BPND anteroventral striatum | 1.68 (0.26) | 1.54 (0.32) | 1.46 (0.47) | 1.60 (0.34)
  [11C]DASB BPND post dorsal caudate | 0.44 (0.15) | 0.35 (0.18) | 0.39 (0.16) | 0.37 (0.19)
  [11C]DASB BPND posterior putamen | 1.36 (0.25) | 1.27 (0.18) | 1.17 (0.39) | 1.32 (0.29)
  [11C]DASB BPND predorsal caudate | 1.08 (0.19) | 0.99 (0.32) | 0.99 (0.34) | 0.98 (0.30)
  [11C]DASB BPND anterior putamen | 1.70 (0.26) | 1.59 (0.26) | 1.49 (0.48) | 1.57 (0.28)
  [11C]DASB BPND midbrain | 2.21 (0.31) | 2.06 (0.30) | 1.98 (0.60) | 2.17 (0.19)
Statistical Analysis 1: Comparison: [11C]DASB Binding Potential Control Women vs [11C]DASB Binding Potential in REC AN vs [11C]DASB Binding Potential in REC ANBN vs [11C]DASB Binding Potential in REC BN; Test type: Superiority; p > 0.05, ANOVA — The p value was calculated and adjusted for multiple comparisons (Bonferroni)

2. Secondary Outcome: Dopamine D2/D3 Receptor Binding as Measured During the PET Scan After Amphetamine Administration
Description: Use PET and [11C]raclopride to explore Dopamine D2/D3 receptor binding potential (BPND) in striatal regions of interest in eating disorder subtypes after amphetamine administration. The Binding Potential (BP) was calculated as BP Non Displaceable (ND) = (VT/VND) -1. [VT = distribution volume in tissue; VND = non-displaceable distribution volume].
Time Frame: 90 min PET scan
Population: Due to technical problems and temporary closure of the PET Facility during the study and consequent lack of time and funding for additional scanning, we were unable to recruit a sufficient number of women recovered from bulimia nervosa (BN) for the AMPHETAMINE CHALLENGE STUDY and therefore no data for this outcome measure were collected in REC BN.
Measure: Mean (Standard Deviation); unit: binding potential (BPND)
Groups:
- [11C]Raclopride Binding Potential Control Women: [11C]raclopride binding potential in control women after amphetamine administration
- [11C]Raclopride Binding Potential in REC AN: [11C]raclopride binding potential in women recovered from restricting type anorexia nervosa (REC AN) after amphetamine administration
- [11C]Raclopride Binding Potential in REC ANBN: [11C]raclopride binding potential in womenrecovered from bulimic type anorexia nervosa (REC ANBN) after amphetamine administration
Arm/Group | [11C]Raclopride Binding Potential Control Women | [11C]Raclopride Binding Potential in REC AN | [11C]Raclopride Binding Potential in REC ANBN
Number analyzed (Participants) | 14 | 13 | 5
binding potential (BPND)
  [11C]raclopride BPND anteroventral striatum | 2.09 (0.22) | 2.01 (0.15) | 1.94 (0.37)
  [11C]raclopride BPND post dorsal caudate | 1.69 (0.27) | 1.62 (0.19) | 1.69 (0.34)
  [11C]raclopride BPND anterior putamen | 2.71 (0.26) | 2.65 (0.22) | 2.60 (0.40)
  [11C]raclopride BPND posterior putamen | 2.53 (0.32) | 2.46 (0.26) | 2.47 (0.40)
  [11C]raclopride BPND predorsal caudate | 2.48 (0.30) | 2.40 (0.14) | 2.47 (0.47)
Statistical Analysis 1: Comparison: [11C]Raclopride Binding Potential Control Women vs [11C]Raclopride Binding Potential in REC AN vs [11C]Raclopride Binding Potential in REC ANBN; A General Linear Model using log([11C]raclopride BPND) after amphetamine administration as dependent variable and Diagnostic Group as independent variable was used. Baseline (before amphetamine administration) [11C]raclopride BPND was used as covariate; Test type: Superiority; p < 0.05, General Linear Model — The p value was calculated and adjusted for multiple comparisons (Bonferroni)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | [11C]Raclopride, [11C]DASB, Amphetamine
All-Cause Mortality (participants affected / at risk) | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 2/85
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | [11C]Raclopride, [11C]DASB, Amphetamine (N=85)
High blood pressure (Cardiac disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT02020408/Prot_SAP_000.pdf